CLINICAL TRIAL: NCT05378802
Title: Comparison of Spontaneous Breathing and Controlled Ventilation
Brief Title: Predict Transpulmonary Pressure Through ZAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Director, Southeast University, China
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ZAM study
Record Dates: First submitted 2021-11-06; First posted 2022-05-18 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Acute Respiratory Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NAVA mode (Experimental): 1. st select a NAVA level that gives peak pressure about 9-10 cm H2O assist keep NAVA level for 15 minutes, do ZAM breaths every 3 minutes (make sure not to disturb the patient). Insp Hold after every ZAM
  2. nd increase NAVA level by 50% and repeat the protocol when patient's breathing has stabilized (only one increase) Do ZAM breaths every 3 minutes (make sure not to disturb the patient). Insp Hold after every ZAM
  Interventions: Other: different modes of mechanical ventilation
- N- PSV mode (Experimental): 1. st PS level of 8-10 cmH2O, keep PS level for 15 minutes, do ZAM every 3 minutes (make sure not to disturb patient). Insp Hold after every ZAM At the end of protocol (minute 15) do one end-inspiratory hold-maneuver and one end-expiratory occlusion.
  2. nd increase PS by 50% and repeat protocol when patient's breathing has stabilized (only 1 increase). Do ZAM every 3 minutes (make sure not to disturb patient). Insp Hold after every ZAM
  Interventions: Other: different modes of mechanical ventilation
- VCV mode (Active Comparator): no spontaneous breathing Set Vt, Ti and RR to match the breathing pattern observed during NAVA. Make sure each change in "level" does not increase the pressure by more than 1 cmH2O.
  Mode PCV no spontaneous breathing-do ZAM after each PS level Increase PSV level from 8 to 20 in steps of 1 cmH2O every 2 minutes. Be careful at the higher pressures.
  Interventions: Other: different modes of mechanical ventilation
- PCV mode (Active Comparator): Increase PSV level from 8 to 20 in steps of 1 cmH2O every 2 minutes. Be careful at the higher pressures The idea is not to have pressures as high as 20 cmH2O, it is important to have high enough VCV & PCV flow rates so we can match the flow rates during spontaneous breathing. You might find that 15 or 16 cmH2O is enough to generate flow rates that match the "maximum" flow rate you saw during spontaneous breathing.
  Interventions: Other: different modes of mechanical ventilation

INTERVENTIONS:
Other: different modes of mechanical ventilation — Four different ventilation modes were performed one by one and respiratory parameters were recorded.

SUMMARY:
Stable patient with ARF spontaneously breathing light sedation (not too awake but with stable breathing pattern) and EAdi >8 uV. Four modes of mechanical ventilation were performed under different support level for the measuring of EAdi, air way pressure and other parameters.

DETAILED DESCRIPTION:
1. Mode NAVA spontaneous breathing select a NAVA level that gives peak pressure about 9-10 cm H2O assist keep NAVA level for 15 minutes, do ZAM breaths every 3 minutes (make sure not to disturb the patient). Insp Hold after every ZAM.

   Increase NAVA level by 50% and repeat the protocol when patient's breathing has stabilized (only one increase).Do ZAM breaths every 3 minutes (make sure not to disturb the patient). Insp Hold after every ZAMAt the end of protocol (minute 15) do one end-inspiratory hold-maneuver and one end-expiratory occlusion.
2. Mode N- PSV spontaneous breathing :PS level of 8-10 cmH2O, keep PS level for 15 minutes, do ZAM every 3 minutes (make sure not to disturb patient). Inspiratory Hold after every ZAM。At the end of protocol (minute 15) do one end-inspiratory hold-maneuver and one end-expiratory occlusion.Increase PS by 50% and repeat protocol when patient's breathing has stabilized (only 1 increase). Do ZAM every 3 minutes (make sure not to disturb patient). Inspiratory Hold after every ZAM.At the end of protocol (minute 15) do one end-inspiratory hold-maneuver and one end-expiratory occlusion.

   Make record of RR, Vt, Flow, Ti during both periods.
3. Mode VCV no spontaneous breathing：Set Vt, Ti and RR to match the breathing pattern observed during NAVA
4. Mode PCV no spontaneous breathing-do ZAM after each PS level：Increase PSV level from 8 to 20 in steps of 1 cmH2O every 2 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Stable patient with acute respiratory failure on invasive mechanical ventilation Can tolerate pressure support ventilation light sedation with RASS between -2 and 1

Exclusion Criteria:

* EAdi<8 uV contraindication for nasogastric tube insertion neuromuscular disease affecting spontaneous breathing lack of informed consent, and patients included in other intervention study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Predicted transpulmonary pressure | 6 hours
  Transpulmonary pressure calculated from airway pressure by Prediction formula

SECONDARY OUTCOMES:
patient-ventilator breath contribution | 6 hours
  An index for quantifying the respective patient and ventilator breath contributions
inspiratory flow | 6 hours
  the inspiratory flow measured by the ventilator

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Qiu, Principal Investigator — Southeast University
Locations (1):
- Zhongda hospital, Southeast university, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
This is a physiological study, we do not intend to disclose the data

REFERENCES:
- [Derived] Liu L, He H, Liang M, Beck J, Sinderby C. Estimation of transpulmonary driving pressure using a lower assist maneuver (LAM) during synchronized ventilation in patients with acute respiratory failure: a physiological study. Intensive Care Med Exp. 2024 Oct 4;12(1):89. doi: 10.1186/s40635-024-00674-z. PMID 39365383